CLINICAL TRIAL: NCT03317522
Title: Maternal Lipids at 28 Weeks Gestation and Offspring Adiposity at Age 5-7 Years in the Hyperglycemia and Adverse Pregnancy Outcome Study
Brief Title: Maternal Lipids and Offspring Adiposity at 5-7 Years
Acronym: HAPO
Status: Completed | Type: Observational
Sponsor: Belfast Health and Social Care Trust (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Diabetes UK (Other)
Responsible Party: Sponsor
Other Study IDs: BelfastHSCT; R01HD034242 (NIH)
Record Dates: First submitted 2017-10-10; First posted 2017-10-23 (Actual); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Adiposity
Keywords: Pregnancy; teratogenesis
MeSH Terms: conditions — Obesity; Teratogenesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples remain for a number of participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Belfast HAPO: All pregnant women who attended the Royal Victoria Maternity Hospital, Belfast were eligible to participate unless they met one or more exclusion criteria.
  All eligible women from the Belfast centre were invited to take part in a prospective observational study involving an additional fasting serum sample for lipids at 28 weeks gestation and long term follow up of their HAPO offspring. Only those women who had remained blinded to oral glucose tolerance test (OGTT) results during pregnancy were included (fasting plasma glucose ≤5·8 mmol/L and 2-hour glucose ≤11·1 mmol/L). Offspring from these pregnancies had anthropometric measurements performed within 72 hours of birth and at age 5-7 years.

SUMMARY:
This study investigates the associations between measured maternal lipids (Total cholesterol, LDL-cholesterol , triglycerides and high-density lipoprotein cholesterol) at 28 weeks' gestation and offspring adiposity at 5-7 years. This was examined in a large observational study based in Belfast, UK.

DETAILED DESCRIPTION:
The concept of fuel mediated teratogenesis, as proposed by Freinkel in his 1980 Banting Lecture, postulated that altered fuel metabolism during pregnancy had a long lasting metabolic effect on the offspring. Although in the intervening years the focus has largely been on maternal glucose as the principal fetal fuel, animal studies have documented that other nutrients such as lipids can also be transferred across the placenta. Furthermore, the latter part of pregnancy is associated with a significant hyperlipidemia including hypercholesterolemia and hypertriglyceridemia. Although the relation of maternal lipids during pregnancy to birth outcomes is well documented, few studies have examined this relation to longer term outcomes. Such an association, if present, would lend further support to the presence of developmental programming in the offspring based on fuel mediated teratogenesis.

Against such a background, the aim of this study was to examine the association between maternal lipids during pregnancy and later offspring adiposity controlled for relevant confounders including maternal body mass index (BMI), gestational glycemia and offspring birth weight.

The Hyperglycemia and Adverse Pregnancy Outcome (HAPO) Study was an international multicentre epidemiologic study that examined the associations of hyperglycemia during pregnancy to adverse maternal/fetal pregnancy outcomes. Eligible pregnant women attended the Royal Victoria Maternity Hospital for an oral glucose tolerance test between 24-32 weeks gestation to assess glucose tolerance. An additional fasting serum sample for analysis of lipids was taken.

The mothers and their offspring were invited to return to the study 5-7 years later. At this visit, offspring weight, height and skin fold thickness measurements were taken.

ELIGIBILITY:
Inclusion Criteria:

* In a pregnant state in the first/second trimester
* Attending the Royal Victoria Maternity Hospital

Exclusion Criteria:

* Age younger than 18 years
* A plan to undergo delivery at another hospital
* An uncertain date of last menstrual period and no ultrasonographic estimation between 6 and 24 weeks of gestational age
* Inability to complete the oral glucose-tolerance test within 32 weeks of gestation
* Multiple pregnancy
* Conception by means of gonadotropin ovulation induction or in vitro fertilization
* Glucose testing before recruitment or a diagnosis of diabetes during the current pregnancy
* Diagnosis of diabetes before the current pregnancy and requiring treatment with medication
* Participation in another study that could interfere with the HAPO study
* Infection with the human immunodeficiency virus or hepatitis B or C virus
* Previous participation in the HAPO study
* Inability to converse in the languages used on centre forms without the aid of an interpreter

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants had to be pregnant to take part in study and therefore only female participants could be selected.
Study Population: All pregnant women who attended the Royal Victoria Maternity Hospital were eligible to participate unless they met one or more of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1224 (Actual)
Dates: Start 2001-01-09 (Actual); Primary Completion 2006-11-04 (Actual); Study Completion 2012-03-14 (Actual)

PRIMARY OUTCOMES:
BMI Z score | 5-7 years
  Adiposity expressed as body mass index (BMI) Z score
Sum of skin fold thicknesses | 5-7 years
  Sum of triceps, subscapular and suprailiac

CONTACTS AND LOCATIONS:
Overall Officials: David R McCance, MD, Principal Investigator — Belfast Health and Social Care Trust

IPD SHARING:
Plan to Share IPD: No